CLINICAL TRIAL: NCT07189221
Title: BUMP2BABY & ME+ (B2B&ME+): A Multi-Country, European Implementation Project to Reduce Adverse Birth Outcomes, Improve Maternal and Child Health and Reduce Non-Communicable Disease Risk
Brief Title: Implementation and Evaluation of Bump2Baby and Me+ Programme for Gestational Diabetes Mellitus in Routine Maternity Care Setting.
Acronym: B2B&ME+
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: National Maternity Hospital, Ireland (Other); Aarhus University Hospital (Other); Liva Healthcare A/S (Unknown); Western Norway University of Applied Sciences (Other); University of Agder (Other); Pomeranian Medical University Szczecin (Other); Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other); Deakin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Bump2Baby and Me+; B2B&ME+ (Other Grant/Funding Number: Health Research Board and Horizon Europe)
Record Dates: First submitted 2025-08-28; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: Pregnancy; GDM; Lifestyle Intervention
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: This study employs a hybrid type 3 implementation-effectiveness design using a non-randomised, ABA intervention approach nested within a longitudinal cohort. The study will compare the delivery of the Monash machine learning GDM screening tool (MMLGST) and mHealth coaching referral during a 3-month intervention block with two 3-month blocks of usual care before and after the intervention. Women identified as being at higher risk of developing GDM using the MMLGST will receive access to the smartphone application that connects them with their health coach, who will provide personalised support about healthy eating, physical activity, mental wellbeing, and infant care from early pregnancy until 9 months after birth. Implementation outcomes will be assessed using the RE-AIM framework, and cost-effectiveness analyses will be conducted from a healthcare system perspective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block A (Usual care phases) (No Intervention): The comparator is usual care (Block A women) as provided at each participating maternity hospital
- Block B (Intervention phase) (Experimental): Women identified as being at risk and likely to benefit from lifestyle intervention will be invited to participate in the B2B&Me+ programme through one of four randomly allocated referral methods (randomisation at site level) that will be rotated every 2 weeks:
  i. Point-of-care (POC) active referral: Women will be directly offered the programme after their appointment, and they will be supported to commence the app sign-up process ii. POC with follow-up phone call: As above plus follow-up call within 48 hours to support enrolment iii. Leaflet with follow-up call: Women will receive an information leaflet about the programme and sign-up process plus a follow-up call within 48 hours to support enrolment iv. Leaflet provided: Women will receive only an information leaflet about the programme and sign-up process
  Interventions: Behavioral: Life Style Intervention

INTERVENTIONS:
Behavioral: Life Style Intervention — The intervention consists of seven related components:
  I. A Bluetooth-enabled weighing scale that syncs with the app to facilitate self-monitoring of weight.
  II. Synchronous coaching sessions conducted on a 1:1 basis between the mHealth coach and participants. There will be 2 synchronous sessions, the first at enrolment and the second between 6-8 weeks postpartum. These sessions typically last 45-50 minutes in length with a follow-up summary video message of the goals discussed and, at the beginning of the mother's journey, the establishing of a change agreement. This is mediated through the live-video feature in the B2B&Me+ mHealth coaching app, but the length and thus number of these sessions is determined by the woman. If the woman is diagnosed with GDM, there will be an opportunity for a third 15-minute synchronous coaching session to review and adjust any lifestyle goals to align with the individual's diabetes management plan.
  III. Asynchronous mHealth coaching that uses a combi
  Arms: Block B (Intervention phase)

SUMMARY:
Gestational diabetes mellitus (GDM) affects approximately 1 in 7 pregnancies globally and is associated with significant short and long-term health consequences for both mothers and infants. While lifestyle interventions during pregnancy can effectively reduce GDM risk and its complications, there is limited guidance on how to translate this evidence into routine antenatal and postpartum care. This project looks to address this gap by exploring the effectiveness of the B2B&Me+ programme within regular maternity services across four European countries and how best to implement it.

Women identified as being at higher risk of developing GDM using a GDM screening tool will receive access to the smartphone application that connects them with their health coach, who will provide personalised support about healthy eating, physical activity, mental wellbeing, and infant care from early pregnancy until 9 months after birth. The participants will be randomised initially to a specific referral pathway for the intervention.

DETAILED DESCRIPTION:
While lifestyle interventions during pregnancy can effectively reduce GDM risk and its complications, there is limited guidance on how to translate this evidence into routine antenatal and postpartum care. Building on the successful Horizon2020-funded Bump2Baby and Me trial, this implementation project seeks to address this gap by testing the real-world effectiveness of the B2B&Me+ programme within regular maternity services across four European countries.

This is a hybrid type 3 implementation-effectiveness study using a non-randomised, ABA intervention design nested within a longitudinal cohort. As a type 3 hybrid, focus is primarily on implementation outcomes while also collecting effectiveness outcomes as they relate to uptake or fidelity of the intervention. The study will compare the delivery of the Monash machine learning GDM screening tool (MMLGDST)12 and mHealth coaching referral during a 3-month intervention block (B) with two 3-month blocks of usual care, before and after the intervention (A blocks).

Block A (Usual care phases): The research staff will briefly explain the data collection aspect of the study and provide an information leaflet. Women will be informed that the study involves collecting anonymised data from their medical records for research purposes, with no additional procedures or interventions beyond their standard care.

Within the intervention block (B), different referral methods will be tested every 2 weeks:

1. Point-of-care (POC) active referral only
2. POC with follow-up phone call
3. Leaflet provided at time of consent with follow-up phone call
4. Leaflet referral only This real-world implementation design will allow us to evaluate not only the clinical effectiveness of the intervention but also the implementation processes, contextual factors, and sustainability of the programme within routine care.

The intervention (B2B&Me+ programme) involved is a lifestyle intervention comprised of the following components:

I. A Bluetooth-enabled weighing scale that syncs with the app to facilitate self-monitoring of weight.

II. Synchronous coaching sessions conducted on a 1:1 basis between the mHealth coach and participants at enrolment and 6-8 weeks postpartum.

III. Asynchronous mHealth coaching that uses a combination of text and video messaging exchanges between the mHealth coach and participant.

IV. Automated push notifications are sent out to participants. V. Participants will receive personalised educational content from their mHealth coach during the asynchronous coaching sessions.

VI. Participants will receive automated push notifications referring to additional content available in the B2B&Me+ app.

VII. Participants will also have access to a virtual social network, through the mHealth coaching app, with other women participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending their first/early antenatal appointments at participating sites
* Gestation less than 24 weeks at enrolment
* Age 18 years or older
* Ability to provide informed consent

Additional for the intervention group (Block B):

* Identified as higher risk for GDM using the MMLGDST
* Ownership of a smartphone compatible with the B2B&Me+ app

Exclusion Criteria:

* 24 weeks gestation or higher
* Multiple pregnancy (twins, triplets, etc.)

Additional for the intervention group (Block B):

* Participation in another health behaviour change intervention study during pregnancy
* Inability to understand the language of the intervention (English in Ireland, Spanish in Spain, Norwegian in Norway, Polish in Poland)
* Severe mental illness, drug or alcohol abuse that would impair ability to participate
* Cancer (not in remission)
* Myocardial infarction in the last three months
* Pre-existing diabetes (Type 1 or Type 2), or early GDM.
* Not owning a smartphone capable of hosting the intervention app

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Penetration and participation rates in early pregnancy GDM screening and intervention | Immediately following intervention.
  The primary analysis will compare penetration across the different blocks (A vs B), participation rates and different referral methods within Block B. This will be analysed using chi-square tests for categorical data and t-tests or ANOVA for continuous data.

SECONDARY OUTCOMES:
Maternal Weight and BMI at baby's birth | At birth of baby.
  Maternal weight (kg) and Body Mass Index (gestational weight gain)
GDM incidence at baby's birth. | At birth of baby
  GDM incidence rate.
Adverse Birth Outcomes | Until birth of last baby included.
  Rates of adverse birth outcomes (pre-eclampsia, preterm birth, birth weight ≥4000g, birth trauma, neonatal respiratory distress, phototherapy, stillbirth/neonatal death, NICU admission or shoulder dystocia, caesarean section/interventions)
Breastfeeding Initiation. | At discharge following birth of baby.
  Breastfeeding initiation rates and on discharge
Healthcare Utilisation. | At birth of baby.
  Healthcare utilisation and costs (hospital stays, specialist consultations)
Maternal weight and BMI at 9 months postpartum | At 9 months postpartum.
  Maternal weight (kg) and Body Mass Index.
Breastfeeding Duration | Up to 9 months postpartum.
  Duration of breastfeeding.
Diet quality | At 9 months postpartum.
  Quality of diet.
Physical Activity | At 9 months postpartum.
  Measure of physical activity.
Implementation Outcomes Evaluated | At 9 months postpartum.
  Evaluation of implementation outcomes per the RE-AIM frame work (Reach, Effectiveness, Adoption, Implementation, Maintenance)

CONTACTS AND LOCATIONS:
Overall Officials: Sharleen O'Reilly, Principal Investigator — University College Dublin

IPD SHARING:
Plan to Share IPD: No